CLINICAL TRIAL: NCT03952416
Title: Patient Engagement Intervention in Inpatient Spinal Cord Injury Rehabilitation
Brief Title: Enhanced Medical Rehabilitation for Spinal Cord Injury
Acronym: EMRSCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Wing Wong, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201803164; NCT05364151 (obsolete NCT alias)
Record Dates: First submitted 2019-05-03; First posted 2019-05-16 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injuries
Keywords: Occupational Therapy; Physical Therapy; Spinal Cord Injury; Patient Engagement; Medical Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Patient Participation

STUDY DESIGN:
Intervention Model Description: Eighty participants with spinal cord injury (SCI) who are admitted to the SCI rehabilitation (at Shirley Ryan Ability Lab) will be split into two groups. This will be randomized. Group 1 will receive the intervention, enhanced medical rehabilitation (EMR) while Group 2 will receive the standard existing rehabilitation, standard of care (SOC).
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants are masked. The care provide and investigator are not mask. Only one research assistant (outcomes assessor) will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (No Intervention): The control group for this study will receive rehabilitation therapy that is recommended and provided by the current healthcare structure. The SOC group will receive therapy only from four therapists who are not trained and supervised in EMR. These therapists will be monitored (videotaped or observed) but will not be not asked to do anything differently with their patients. The investigators recognize that spillover of therapist EMR training to untrained therapists is a concern. Thus, the investigators will ask therapists in the EMR group to agree not to share any of the training with non-trained therapists over the course of the study, and the investigators will provide free EMR training to the non-trained therapists once the treatment phase of the study is complete.
- Enhanced Medical Rehabilitation (EMR) (Experimental): Patients in the EMR group will also receive the recommended rehabilitation therapy, but they will receive therapy only from four therapists who are trained and supervised in EMR. The therapy sessions will follow EMR protocol. EMR is a set of behavioral skills that therapists can incorporate into their daily therapy sessions to increase patient engagement and achieve a high intensity of therapy, thereby improving functional and psychosocial outcomes of patients in medical rehabilitation.
  Interventions: Behavioral: Enhanced Medical Rehabilitation (EMR)

INTERVENTIONS:
Behavioral: Enhanced Medical Rehabilitation (EMR) — EMR is a set of behavioral skills that therapists can incorporate into their daily therapy sessions to increase patient engagement and achieve a high intensity of therapy, thereby improving functional and psychosocial outcomes of patients in medical rehabilitation. EMR was built on theories of behavior change, including social cognitive theory and self-regulatory theory, and their applications to patient engagement, such as the Health Action Process Approach and motivational interviewing. It has three foci: (1) a patient-directed, interactive approach stemming from patient-centered goals ("Patient as boss"); (2) frequent feedback to patients on their efforts and progress ("Link activities to personal goals"); and (3) increased rehabilitation intensity ("Optimize intensity").
  Arms: Enhanced Medical Rehabilitation (EMR)

SUMMARY:
Background: Patient engagement is a cornerstone of patient-centered care. Studies show that an increased level of patient engagement in medical rehabilitation is associated with greater functional recovery. To achieve higher levels of patient engagement, it is important to improve therapists' techniques for goal setting and clinician-therapist communication. Thus, we have developed a manualized intervention for post-acute rehabilitation, Enhanced Medical Rehabilitation (EMR), which is an evidence-based program to increase patient engagement and achieve a greater intensity of therapy, thereby optimizing the patient's functional and psychosocial recovery. EMR is an integrated set of skills for occupational and physical therapists that transform rehabilitation through (1) a patient-directed, interactive approach; (2) increased treatment intensity; and (3) frequent feedback to patients on effort and progress. We have developed training and supervision methods to enable therapists to carry out these skills with high fidelity. In our previous EMR study of older adults in skilled nursing facilities, patients treated by EMR-trained therapists had greater engagement in therapy, higher-intensity therapy sessions, and better functional outcomes. Due to the complexity of the inpatient spinal cord injury (SCI) rehabilitation environment, it is unknown whether the EMR program will be clinically relevant to inpatient rehabilitation settings and acceptable to SCI populations. Therefore, it is necessary to conduct a systematic adaptation approach to address all hospital- and provider-level barriers, and test this adapted program to a new setting (inpatient rehabilitation) and a new population (patients with SCI), without compromising the core elements of the original EMR.

Objective: We propose to adopt the EMR program for use in inpatient SCI rehabilitation settings using an implementation science-driven approach. We also propose a randomized trial of 80 patients with SCI to test the effects of EMR on improving engagement and treatment intensity, as well as functional and psychosocial outcomes over standard of care (SOC) rehabilitation.

Methods: We will randomize patients into EMR or SOC groups. For the EMR group, four therapists will be trained and supervised in EMR and will incorporate EMR techniques into therapy sessions. In the SOC group, four therapists will carry out therapy sessions as usual.

Expected Outcomes: With respect to EMR intervention adaptions, we hypothesize that the EMR program, including a treatment manual and other materials, will be customized with input from our Spinal Cord Injury-Community Advisory Board (SCI-CAB). Patients randomized to EMR will have greater engagement and intensity and greater functional and psychosocial recovery compared to those randomized to SOC rehabilitation.

Significance: The impact is high. EMR is patient-centered rehabilitation, and it is designed for real-world clinical practice. Success in this line of research will improve therapists' skills working with patients and optimizing patient outcomes, ensuring that inpatient SCI rehabilitation is more patient-centered, to the benefit of individuals with SCI.

DETAILED DESCRIPTION:
Patient engagement (or participation) is a critical cornerstone for patient-centered care, including inpatient spinal cord injury (SCI) rehabilitation. Researchers have defined patient engagement as a deliberate effort and commitment to working toward the goals of rehabilitation therapy, typically demonstrated through active participation and cooperation with treatment providers. Our previous work has shown that patient engagement is an important determinant of positive rehabilitation outcomes, as higher levels of patient engagement are associated with increased functional improvement and shorter lengths of stay. In the field of SCI research, we recently investigated personalized trajectories of engagement in occupational therapy (OT) inpatient rehabilitation in relation to patient outcomes. We found that a subgroup of patients who sustained high levels of engagement during the rehabilitation stay were more likely to have better functional, psychosocial, and participation outcomes at discharge and one-year post-injury than subgroups of patients whose levels of engagement progressively deteriorated. Other researchers found similar results for physical therapy (PT) inpatient interventions, suggesting that engagement in rehabilitation is predictive of whether the patient is discharged to home and the patient's level of involvement in work or school one-year post-injury. Given the promising results of Enhanced Medical Rehabilitation (EMR) interventions in SNFs, an important step for expanding the use of EMR is to customize it to other target populations and practice settings in order to enhance its reach. We propose a modification of EMR adapted for inpatient SCI rehabilitation using the Collaborative Intervention Planning Framework. We will then pilot test the efficacy of EMR versus SOC rehabilitation on improving patient engagement and treatment intensity (processes), and enhancing function and psychosocial recovery (outcomes). Thus, the aims of this study are to conduct intervention adaptations to the EMR program for patients in inpatient SCI rehabilitation and conduct a pilot RCT to demonstrate the benefits of EMR over SOC treatment in inpatient SCI rehabilitation.

Despite the demonstrated relationship between patient engagement and functional outcomes/psychosocial recovery, several factors may affect engagement in rehabilitation, including goal setting, therapeutic connection, personalization, patient-centered rehabilitation, autonomy, and feedback. Many of these factors are influenced by how therapists deliver their interventions; the patient-clinician interaction is the foundation for successful engagement in rehabilitation. Thus, achieving strong patient engagement depends on a high level of targeted interaction from therapists responsible for providing rehabilitation services. Unfortunately, improving the therapist's ability to engage patients during clinical practice is challenging given the changing and competing demands of the real-world rehabilitation environment. This "environmental barrier" concurs with findings from our recent qualitative study exploring perceived barriers of patient engagement implementation in SCI rehabilitation. We found that unavailability of hospital resources and insurance restrictions can undermine rehabilitation by restricting the patient's ability to reach personal treatment goals. For instance, one patient discussed treatment goals that may not be person-centered, but rather are centered on satisfying insurance reimbursement: "They [providers] create goals. They have to. It's part of the insurance thing. They have to report every couple of weeks to see where you are going, how you are progressing against something measurable, I understand that. The problem is you get folks [therapists who say] 'Oh I got to write some goals for this guy. Oh, well, he will be able to pick his nose.'" Similarly, another hospital-level barrier that undermines engagement in SCI rehabilitation is the lack of structured training for therapists to support patient engagement. A therapist in the focus group said, "I mean…[the] individual manager, the team leader will find a way to foster staff development to help with engagement. I can't think of any such big hospital-wide initiatives." To address these barriers, we developed Enhanced Medical Rehabilitation (EMR) to teach occupational and physical therapists a set of behavioral skills to engage patients and involve them in high-intensity therapy in order to optimize functional and psychosocial outcomes of patients in medical rehabilitation (please refer to Research Plan for details on EMR). It is important to note that EMR is a "how" intervention, not a "what" intervention. Its skill set integrates into existing OT/PT practices rather than adding new activities, exercises, or another specialist to the setting. The difference between EMR and standard of care (SOC) OT/PT is the effort necessary to engage the patient and provide high-intensity therapy. For this reason, EMR can integrate well into real-world OT/PT practices regardless of the patient's primary impairment, comorbidities, or other contextual factors. Currently, we have successfully tested EMR for older adults receiving post-acute rehabilitation. In particular, we found that: (1) EMR can be implemented in real-world skilled nursing facilities (SNFs). Occupational and physical therapists who were trained and supervised carried out EMR with high treatment fidelity. (2) Patients receiving services from EMR therapists demonstrated greater treatment intensity and patient engagement in rehabilitation compared to those receiving services from SOC therapists. (3) EMR improves rehabilitation outcomes. Patients randomized to EMR had better improvement in depressive symptoms and function than controls. (4) EMR overcomes barriers to rehabilitation. Those vulnerable to poor rehabilitation outcomes-patients with multiple medical comorbidities, cognitive impairment, and/or depression-benefitted the most from EMR. In spite of preliminary evidence suggesting the benefits of EMR, it remains unknown whether the EMR skills, therapist training, and coaching protocol, treatment fidelity methods, processes, and outcome measures developed for older adults in SNFs will be clinically relevant to the inpatient rehabilitation setting and acceptable to SCI populations. Thus, we will utilize an established implementation science approach to customize an existing EMR program to a new patient population and a new setting. We will use the Collaborative Intervention Planning Framework (CIPF) to customize the EMR program to patients with SCI in inpatient rehabilitation facilities (IRFs). This framework will help us move from intervention planning to pilot test through a randomized controlled trial (RCT) to assess the feasibility of the adapted EMR and explore its initial effects.

This proposed study addresses the problem of suboptimal patient engagement in SCI rehabilitation. Most persons following SCI go to an IRF for an average of 35 days of OT/PT. This is a narrow window of opportunity for persons with SCI to regain enough function to return home and live independently. Unfortunately, "failed rehabilitation" often results because SOC therapy is not sufficiently patient centered and is of low intensity. As a result, SOC therapy does not adequately engage and benefit patients for positive rehabilitation outcomes.

Post-acute OT/PT is often low in intensity. This observation may seem counterintuitive, as IRF rehabilitation involves up to three hours of daily contact. However, actual time spent on OT/PT is typically less than that. Scheduled therapy time may greatly overestimate actual active time during sessions; studies using ACTi Graph accelerometry monitors and observers counting repetitions have found a low intensity of treatment in a variety of post-acute rehabilitation settings. Two major factors may account for this low intensity of post-acute rehabilitation. First, occupational and physical therapists often do not strive for high intensity. Second, the interaction with patients may be unengaging for patients because therapists do not explicitly use principles of engagement, including patient-directed therapy and frequency feedback. The low intensity of post-acute rehabilitation has caught the attention of rehabilitation providers and policymakers, with evidence showing that rehabilitation outcomes have not significantly improved despite an increase in billed therapy hours over recent decades.

Research shows a positive relationship between patient engagement and rehabilitation outcomes. Thus, to improve the outcomes of patients in inpatient SCI rehabilitation, we must address the problems of low intensity and poor patient engagement in rehabilitation. EMR is an evidence-based intervention that therapists can use to engage patients participating in high-intensity therapy and that has been successfully tested in SNFs. Yet, to date, there is no data showing that EMR can work in inpatient SCI rehabilitation facilities. Thus, the overall goals of this project are to adapt the EMR intervention to a new patient population (i.e., from older adults to SCI) and new setting (i.e., from SNFs to IRFs), as well as to assess the feasibility of this adapted intervention to improve functional and psychosocial outcomes of inpatients with SCI. If we demonstrate the feasibility and efficacy of adapted EMR, our next step is to conduct a full-scale test of the effectiveness of the adapted EMR and its implementation in inpatient SCI rehabilitation settings. Success in this line of research will ultimately improve inpatient SCI rehabilitation, making it more patient centered, to benefit the 285,000 people currently living with SCI, people with a new injury, and their families.

This application is consistent with the Foundation's mission to improve the quality of life for those affected by and living with SCI. Our study aims to develop an evidence-based intervention that teaches therapists a set of patient engagement skills with the goal of improving patient function and other rehabilitation outcomes. This intervention will establish a new standard for the delivery of SCI care, particularly in the area of rehabilitation. We propose that therapists who acquire EMR skills will improve patients' engagement and the intensity of therapy, leading to better function, treatment satisfaction, and life satisfaction, and reduce depressive symptoms. Additionally, this EMR project will support the Foundation's core value of psychosocial research to inform best practices that are more patient centered by optimizing quality interactions between practitioners and individuals with SCI.

AIM 1: Conduct intervention adaptations to the EMR program for patients in inpatient SCI rehabilitation Aim 1.1: Create a stage to foster partnership and collaboration among implementers of the EMR program Hypothesis 1.1: An SCI Community Advisory Board (SCI-CAB), including clinicians, administrators, investigators, and peer specialists/patient advocates, will be assembled to learn and review the EMR program.

Aim 1.2: Conduct needs assessment to understand the problems of current SCI practice Hypothesis 1.2: SCI-CAB members will successfully identify the engagement-related needs and areas for intervention adaptations for inpatients with SCI.

Aim 1.3: Review intervention components of the original EMR program to identify targets for adaptation Hypothesis 1.3: SCI-CAB members will successfully identify specific adaptations to intervention content or delivery, including the objectives, methods, materials, and theoretical foundations of the EMR program.

Aim 1.4: Incorporate adaptations into the EMR program for inpatient SCI rehabilitation Hypothesis 1.4: We will finalize the EMR manual and materials, and train EMR supervisor and therapists.

AIM 2: Conduct a pilot RCT to demonstrate the benefits of EMR over SOC treatment in inpatient SCI rehabilitation Aim 2.1: Examine the preliminary efficacy of EMR for improving patient engagement and treatment intensity Hypothesis 2.1: EMR will improve engagement and intensity to a greater extent than SOC rehabilitation.

Aim 2.2: Examine the preliminary efficacy of EMR for improving functional and psychosocial outcomes Hypothesis 2.2: EMR will improve functional and psychosocial outcomes to a greater extent than SOC rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* (1) inpatient therapists specializing in SCI patients for at least six months
* (2) practicing on one of two SCI units at the SRAL
* (3) willing to collect study measures
* (4) willing to be videotaped for therapy sessions with patients
* (5) willing and able to participate in EMR training and supervision sessions.

Exclusion Criteria:

* (1) inpatient therapists specializing in SCI for less than six months
* (2) not willing/able to follow study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Function: CARE Tool | 1 Month
  The investigators will use the CARE tool to measure the level of independence as the primary outcome at both admission and discharge.
  At admission, the investigators will use the CARE tool to measure the patient's independence before the treatment. At discharge, the investigators will use the same CARE tool to measure the patient's independence after the treatment. This clinician-rated measure contains 18 items composed of 13 motor and 5 cognitive tasks. Tasks are rated on a 6-point ordinal scale that ranges from the minimum score of 1 (dependent) to a maximum score of 6 (independence). A higher score indicates greater independence. The investigators will use CARE mobility and self-care scores to reflect patient's ability to perform mobility and self-care tasks, respectively.

SECONDARY OUTCOMES:
Life Satisfaction: Satisfaction with Life Scale | 1 Month
  The investigators will use the Satisfaction with Life Scale to measure the psychological functioning as the secondary outcome. This measure will be measured at both admission and discharge of inpatient rehabilitation.
  At admission, the investigators will use the Satisfaction with Life Scale to measure the patient's psychological functioning before the treatment. At discharge, the investigators will use the same Satisfaction with Life Scale to measure the patient's psychological functioning after the treatment. This self-report measure contains a single item assessing overall life satisfaction, along with eight additional items that are domain specific (e.g., self-care, vocational situation). Items are answered on a 6-point scale that ranges from 1 (very dissatisfied) to 6 (very satisfied). A higher score indicates greater life satisfaction. It has been tested and validated in SCI, with adequate internal consistency of items (α = 0.95).
Depression: Patient Health Questionnaire-9 | 1 Month
  A measure of psychosocial recovery; this self-report measure assesses the presence and intensity of depressive symptoms. It contains 9 questions rated based on the frequency of occurrence of symptoms in the past 2 weeks (from 0 = "Not at all" to 3 = "Nearly every day"). A higher score indicates greater symptomatology. PHQ-9 has been shown as a promising tool to identify probable major depressive disorder (MDD) in people with SCI.

CONTACTS AND LOCATIONS:
Overall Officials: Piper Hansen, OTD, Study Director — Shirley Ryan Ability Lab
Locations (1):
- Shirley Ryan Ability Lab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.